CLINICAL TRIAL: NCT05317273
Title: Incidence and Risk Factors of Urosepsis in Patients With Urinary Tract Calculi Receiving Surgical Intervention
Brief Title: Urosepsis in Patients With Urinary Tract Calculi Receiving Surgical Intervention
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Aphichat Suphathamwit,, Assistant Professor, Mahidol University
Other Study IDs: 2022_1
Record Dates: First submitted 2022-03-20; First posted 2022-04-07 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Urosepsis; Urinary Tract Stone
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Urosepsis is one of major cause of the overall sepsis leading to high morbidity and mortality, which commonly resulted from urinary tract calculi. The investigator aim to identified the incidence and risk factors of urosepsis in the patients with urinary tract calculi underwent surgical intervention in tertiary-care university hospital.

DETAILED DESCRIPTION:
Sepsis is one of the leading cause of death of hospitalized patients in Thailand. Urosepsis or sepsis which originate from urinary tract infection was reported around 9-31% of the overall sepsis syndrome. Urinary tract calculi requiring surgical procedure was reported as a common cause of urinary tract infection. Therefore, the investigators aimed to identified the incidence and risk factors of urosepsis in the patients with urinary tract calculi underwent surgical intervention in tertiary-care university hospital.

Moreover, the patients with sepsis syndrome will be suffered from many complications such as acute respiratory distress syndrome, acute kidney injury, etc. Currently, there were many early waring scores to predict the risk of complications to help promptly treatment and decrease the severity. The investigator would like to compare the systemic inflammatory response syndrome (SIRS) criteria,Modified Early Warning Score (MEWS) and Quick Sequential Organ Failure Assessment (qSOFA) score to the prediction of postoperative complications in this group of patients.

The last primary objective of this study is to follow the course of the patients diagnosed as urosepsis if they had been treated properly according to the sepsis bundle guideline and their outcome.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients with urinary tract calculi requiring surgical procedure

Exclusion Criteria:

- Incomplete data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with urinary tract calculi requiring surgical procedure; percutaneous nephro-ureterolithotrypsy (PCNL), Retrograde intrarenal surgery (RIRS), Ureteroscopic lithotrypsy (URSL) and open lithotomy in tertiary-care university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 865 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Rate of urosepsis diagnosis | 7 days after surgery
  According to urine exam and SIRS criteria of sepsis
Date of urosepsis diagnosis | 7 days after surgery
  date of diagnosis of urosepsis
Mortality rate | 30 days after surgery
  Number of deceased patient after surgery

SECONDARY OUTCOMES:
Length of stay | 7 days after surgery
  * hospital stay
  * intensive care unit stay
Rate of intensive care unit admission | 7 days after surgery
  Number of patients required ICU admission
Rate of blood transfusion | 7 days after surgery
  Amount of blood transfusion in unit during admission
Rate of mechanical ventilation requirement | 7 days after surgery
  Number of patient required mechanical ventilation support
Rate of re-operation | 7 days after surgery
  Number of patients require second procedure at the same admission
Prevalence of acute kidney injury | 30 days after surgery
  According to KDIGO criteria
Rate of renal replacement therapy requirement | 30 days after surgery
  Number of patients require renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Aphichat Suphathamwit, M.D., Principal Investigator — Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University, THAILAND
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Southern JB, Higgins AM, Young AJ, Kost KA, Schreiter BR, Clifton M, Fulmer BR, Garg T. Risk Factors for Postoperative Fever and Systemic Inflammatory Response Syndrome After Ureteroscopy for Stone Disease. J Endourol. 2019 Jul;33(7):516-522. doi: 10.1089/end.2018.0789. Epub 2019 Jan 22. PMID 30569755
- [Background] Blackmur JP, Maitra NU, Marri RR, Housami F, Malki M, McIlhenny C. Analysis of Factors' Association with Risk of Postoperative Urosepsis in Patients Undergoing Ureteroscopy for Treatment of Stone Disease. J Endourol. 2016 Sep;30(9):963-9. doi: 10.1089/end.2016.0300. Epub 2016 Jul 13. PMID 27317017
- [Background] Amier Y, Zhang Y, Zhang J, Yao W, Wang S, Wei C, Yu X. Analysis of Preoperative Risk Factors for Postoperative Urosepsis After Mini-Percutaneous Nephrolithotomy in Patients with Large Kidney Stones. J Endourol. 2022 Mar;36(3):292-297. doi: 10.1089/end.2021.0406. PMID 34569289
- [Background] Grosso AA, Sessa F, Campi R, Viola L, Polverino P, Crisci A, Salvi M, Liatsikos E, Feu OA, DI Maida F, Tellini R, Traxer O, Cocci A, Mari A, Fiori C, Porpiglia F, Carini M, Tuccio A, Minervini A. Intraoperative and postoperative surgical complications after ureteroscopy, retrograde intrarenal surgery, and percutaneous nephrolithotomy: a systematic review. Minerva Urol Nephrol. 2021 Jun;73(3):309-332. doi: 10.23736/S2724-6051.21.04294-4. Epub 2021 Apr 22. PMID 33887891
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Churpek MM, Snyder A, Han X, Sokol S, Pettit N, Howell MD, Edelson DP. Quick Sepsis-related Organ Failure Assessment, Systemic Inflammatory Response Syndrome, and Early Warning Scores for Detecting Clinical Deterioration in Infected Patients outside the Intensive Care Unit. Am J Respir Crit Care Med. 2017 Apr 1;195(7):906-911. doi: 10.1164/rccm.201604-0854OC. PMID 27649072
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542